CLINICAL TRIAL: NCT02020915
Title: Ultrasound Guided Lateral Sphincterotomy: Long Term Results
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Michael Sørensen, Consultant, Hvidovre University Hospital
Other Study IDs: Sphincterotomy MSOE
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Focus: Anal Incontinence After Lateral Sphincterotomy for Chronic Anal Fissure
MeSH Terms: interventions — Lateral Internal Sphincterotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic anal fissure: Patients are included who had previous treatment with diltiazem or glycerol-nitrate and botox injections
  Interventions: Procedure: lateral sphincterotomy; Procedure: ultrasound guided lateral sphincterotomy

INTERVENTIONS:
Procedure: lateral sphincterotomy
Procedure: ultrasound guided lateral sphincterotomy

SUMMARY:
Ultrasound guided placement of the knife intersphincteric increases accuracy and safety during sphincterotomy. Secondly 3-D ultrasound visualizes that the internal anal sphincter is divided.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing lateral sphincterotomy for chronic anal fissure

Exclusion Criteria:

* Previous diltiazem treatment og botox injections were not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lateral sphincterotomy for chronic anal fissure
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2007-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Anal incontinence | 5 years or more

SECONDARY OUTCOMES:
Healing of fissure | 5 years or more

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark